CLINICAL TRIAL: NCT05641194
Title: EaseAlert: Tactile Firefighter Alerting System Designed to Reduce Negative Cardiovascular Outcomes and Sleep Disturbances
Brief Title: EaseAlert: Tactile Firefighter Alerting System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Embry-Riddle Aeronautical University (Other)
Collaborators: National Development and Research Institutes, Inc. (Other)
Responsible Party: Principal Investigator, Joel Billings, Ph.D., Assistant Professor, Embry-Riddle Aeronautical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 22-131
Record Dates: First submitted 2022-10-28; First posted 2022-12-07 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Heart Rate; Sleep Habit; Sleep

STUDY DESIGN:
Intervention Model Description: 1. Legacy Alerting System Description: Standard alerting system in place at the fire station.
  2. Intervention 2: EaseAlert Standalone Description: EaseAlert will activate and alert the subject of an emergency call without the legacy alerting system. EaseAlert (standalone) replaces the legacy alerting system.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm - intervention (Experimental)
  Interventions: Device: Legacy Alerting System; Device: Intervention 2: EaseAlert Standalone

INTERVENTIONS:
Device: Legacy Alerting System — Description: Standard alerting system in place at the fire station.
Device: Intervention 2: EaseAlert Standalone — Description: EaseAlert will activate and alert the subject of an emergency call without the legacy alerting system. EaseAlert (standalone) replaces the legacy alerting system.

SUMMARY:
The purpose of this research is to test a commercially viable Fire Fighter Altering System (FFAS) comprised of proprietary wearables and optional bed shakers called BunkAlerts; collectively "personal alerting devices" as an alternative approach to the traditional fire alarm system used in fire stations. Participants (fire fighters) will be asked to take part in the study to investigate the impact of the new FFAS on cardiovascular response and sleep. This study includes three phases: 1) baseline, 2) implementation of EaseAlert FFAS with traditional alarm, and 3) implementation of EaseAlert FFAS without traditional alarm. Participants will be asked to wear an Actigraph wGT3x-BT and Polar H10 device to record sleep and heart rate data for 12 days at work in addition to EaseAlert FFAS device for 8 out of the 12 days at work. They will also be asked to complete a questionnaire and complete daily journal entries.

DETAILED DESCRIPTION:
Sudden cardiac death (SCD) has been the leading cause of on-duty death (ODD) in the fire service over the past several decades, accounting for 51.6% of all ODDs in 2019. The primary factors that contribute to SCD among firefighters are overexertion and stress, and SCD is most likely to occur during fire suppression and alarm response. When an emergency occurs, firefighters are alerted/awoken by loud mechanical bells. This high noise level may induce a stress response triggering a cardiovascular event. In fact, "high levels of environmental noise fuel cardiac risk" by stimulating the amygdala and inflaming the arteries. While other companies have attempted to modernize alerting systems, they failed to address the problem of stressful alarms because they focus on alerting "stations" not individual firefighters. A significant need exists to develop a less stressful alerting system for firefighters. The objective of this SBIR Phase I R43 research study is to develop a commercially viable Fire Fighter Alerting System (FFAS) comprised of proprietary wearables and optional bed shakers called BunkAlerts. Collectively "personal alerting devices," the wearables and BunkAlerts enhance the alerting process for firefighters by replacing jarring audible alarms with tactile alerts delivered to the firefighter's wrist. This alternative approach is designed to significantly decrease tachycardic responses associated with legacy alerting systems. Meeting this need has the potential to reduce firefighter ODDs and improve the quality of life for the 15.4 million firefighters around the world. The feasibility of EaseAlert's FFAS is reinforced by preliminary data collected during field testing with six (6) fire departments in three (3) states where EaseAlert's prototype FFAS ("Gen 1") successfully delivered over 10,000 alerts to firefighters called to an emergency with no calls missed. The potential for the FFAS to reduce stress and SCD risk among firefighters is supported by preliminary data which shows that: 1) noise triggers a startle response and 2) tactile alerts are associated with positive valence and high arousal. The proposed research will be accomplished with two aims: Aim 1 - develop a commercially viable FFAS and Aim 2 - determine the effectiveness of the FFAS in reducing cardiac reactivity and improving sleep. EaseAlert will leverage the Gen 1 FFAS as a foundation for developing its Gen 2 FFAS outlined in Aim 1. Aim 2 will test two study hypotheses in a within-subjects pilot clinical trial design: (H2.1) that EaseAlert will result in a significant reduction in the stress response to alarms compared to traditional auditory alerting systems, and (H2.2) EaseAlert will result in a significant improvement in sleep efficiency.

ELIGIBILITY:
Inclusion Criteria:

-

Participants must meet the following inclusion criteria:

* Firefighters must be willing participants be over the age of 18 years
* Have worked at their department for a minimum of two months (career department only) so that circadian rhythm is adjusted to the schedule
* No extended absence or shift trading among the firefighters foreseen during the trial.
* Nighttime call/run volume averaging at least one emergency call
* Interest among the crew members to participate in the trial

Inclusion criteria for departments will include, but not be limited to:

* Willingness to participate by department's chief and/or his/her designee
* No past experience with the EaseAlert FFAS
* Four or more firehouses/stations
* Willingness to identify a departmental point of contact for collaboration with the research team
* Interest among crews to test the new alert system.

Exclusion Criteria:

* non firefighter

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2023-08-26 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Heart Rate (mean) | Change from baseline Heart Rate to post interventions (6 days from baseline). Outcome will be assessed over 1 day per intervention.
  Heart Rate will be measured with Polar H10 Heart Rate Chest Strap Monitor connected via Bluetooth to wGT3X-BT Actigraphy device. Change from baseline Heart Rate to post interventions
Heart Rate (max) | Change from baseline Heart Rate to post interventions (6 days from baseline). Outcome will be assessed over 1 day per intervention.
  Heart Rate will be measured with Polar H10 Heart Rate Chest Strap Monitor connected via Bluetooth to wGT3X-BT Actigraphy device. Change from baseline Heart Rate to post interventions. Max HR will factor subjects' age.
Sleep Efficiency | Change from baseline to post interventions (6 days from baseline). Outcome will be assessed over 1 day per intervention.
  Sleep Efficiency will be measures by wrist actigraphy (device: wGT3X-BT). Actilife 6.0 (issued by ActiGraph Co.) will be used to analyze actigraphy data. Sleep Efficiency is calculated by dividing (total sleep time by total time in bed) X 100. Change from baseline sleep efficiency to post interventions.

SECONDARY OUTCOMES:
Satisfaction with EaseAlert during Night | Change from baseline night satisfaction to post interventions (6 days from baseline). Outcome will be assessed over 1 day per intervention.
  Satisfaction with EaseAlert during the night will be assessed with a 10-point VAS Likert scale (lower scores indicate worse outcome) and an open ended option for additional thoughts. Change from baseline night satisfaction to post interventions.
Satisfaction with EaseAlert during Day | Change from baseline day satisfaction to post interventions (6 days from baseline). Outcome will be assessed over 1 day per intervention.
  Satisfaction with EaseAlert during the day will be assessed with a 10-point VAS Likert scale (lower scores indicate worse outcome) and an open ended option for additional thoughts. Change from baseline day satisfaction to post interventions.
Pre-bed anxiety/stress | Change from baseline pre-bed anxiety/stress to post interventions (6 days from baseline). Outcome will be assessed over 1 day per intervention.
  Pre-bed anxiety/stress will be assessed with a 10-point VAS Likert scale (higher scores indicate worse outcomes) prior to bed. Change from baseline pre-bed anxiety/stress to post interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Joel M Billings, Ph.D., Principal Investigator — Embry-Riddle Aeronautical University
Locations (2):
- United States (2):
  - Central Jackson County Fire District, Blue Springs, Missouri
  - Stillwater Fire Department, Stillwater, Oklahoma

IPD SHARING:
Plan to Share IPD: No